CLINICAL TRIAL: NCT01063478
Title: A Phase I Dose Escalation Study of RAD001 in Combination With Chemotherapy and Radiation in Patients With NSCLC
Brief Title: Dose Escalation Study of RAD001 in Combination w/Chemotherapy & Radiation in Patients With NSCLC
Acronym: RAD001
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Poor accrual
Sponsor: University of Chicago (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09-384-B
Record Dates: First submitted 2010-02-03; First posted 2010-02-05 (Estimated); Last update posted 2014-01-17 (Estimated); Status verified 2014-01

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: Non-Small Cell; Lung Cancer; Unresectable advanced NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — Everolimus; Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- RAD001, Chemotherapy, Radiation (Experimental): RAD001 + Chemotherapy and Radiation
  Interventions: Drug: RAD001 (in addition to standard radiation and chemotherapy)

INTERVENTIONS:
Drug: RAD001 (in addition to standard radiation and chemotherapy) — Standard radiation and chemotherapy (cisplatin and pemetrexed) + RAD001
  Other Names: RAD001 (Everolimus)

SUMMARY:
The purpose of this study is to understand the effects (good and/or bad) of the addition of RAD001 to standard radiation and chemotherapy (cisplatin and pemetrexed) for patients with non-small cell lung cancer.

DETAILED DESCRIPTION:
In oncology, clinical experience with RAD001 has been based on a number of phase I and II studies with single agent RAD001 as well as phase Ib and II studies of RAD001 in combination with other chemotherapeutic and molecular targeted agents, including paclitaxel, gemcitabine, and erlotinib among others. More recently, a phase III trial of single agent RAD001 in patients with metastatic renal cell carcinoma who had failed therapy with VEGF tyrosine kinase inhibitors was completed. Clinical experience for indications other than oncology comes from single dose studies in healthy volunteers, and studies in solid organ transplant patients, where RAD001 was administered with other immunosuppressive agents.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed NSCLC of any type
* Disease stage. Patients with unresectable stage II, stage III, and Mx are eligible. This includes patients who are being considered as surgical candidates after induction chemoradiation. Patients with Mx or M1 disease whose life-span and prognosis are felt to be dominated by the locoregional disease in the chest and are candidates for chemoradiotherapy are also eligible.
* Patients with pleural effusion that is transudative, cytologically negative and non- bloody are eligible if the radiation oncologist feels that the tumor can be encompassed within a reasonable field of radiotherapy.
* If a pleural effusion is of such a small size that a thoracentesis is not possible, then the patient is eligible
* Patients with malignant pleural or pericardial effusions are not eligible
* Patients will be eligible with or without measurable or evaluable disease. Patients with both measurable and evaluable disease will be evaluated for criteria for measurable disease
* Measurable disease is defined according to RECIST criteria
* Evaluable disease is defined as lesions apparent on CT which do not fit criteria for measurability.
* Ill defined masses associated with post obstructive changes
* Mediastinal or hilar adenopathy measurable in only one dimension
* Age ≥ 18 years
* ECOG performance status ≤ 2
* Life expectancy > 6 months
* Adequate lung function as defined by an 02 saturation that is ≥ 90% on room air
* Adequate bone marrow function as shown by: ANC ≥ 1.5 x 109/L, Platelets ≥ 100 x 109/L, Hb >9 g/dL Adequate liver function as shown by: serum bilirubin ≤ 1.5 x ULN, ALT and AST ≤ 2.5x ULN (≤ 5x ULN in patients with liver metastases), INR and PTT ≤1.5. (Anticoagulation is allowed if target INR ≤ 1.5 on a stable dose of warfarin or on a stable dose of LMW heparin for >2 weeks at time of randomization.)
* Adequate renal function: serum creatinine ≤ 1.5 x ULN
* Fasting serum cholesterol ≤300 mg/dL OR ≤7.75 mmol/L AND fasting triglycerides ≤ 2.5 x ULN. NOTE: In case one or both of these thresholds are exceeded, the patient can only be included after initiation of appropriate lipid lowering medication.
* Informed consent must be obtained from all patients prior to beginning therapy. Patients should have the ability to understand and the willingness to sign a written informed consent document.
* Radiation therapy requirements: Patient must have a completed treatment plan approved by the protocol review team

Exclusion Criteria:

* Patients who have received prior radiation or chemotherapy for the current diagnosis of NSCLC (patients who received surgery only for a prior NSCLC are eligible if the current diagnosis is felt to represent a new primary, and the PFT's would allow for concurrent chemoradiation)
* Patients, who have had a major surgery or significant traumatic injury within 4 weeks of start of study drug, patients who have not recovered from the side effects of any major surgery (defined as requiring general anesthesia) or patients that may require major surgery during the course of the study
* Prior treatment with any investigational drug within the preceding 4 weeks
* Patients receiving chronic, systemic treatment with corticosteroids or another immunosuppressive agent. Topical or inhaled corticosteroids are allowed.
* Patients should not receive immunization with attenuated live vaccines within one week of study entry or during study period
* Other malignancies within the past 3 years except for adequately treated carcinoma of the cervix, basal or squamous cell carcinomas of the skin, or breast DCIS, who may be included if the diagnosis was within 3 years.
* Patients who have any severe and/or uncontrolled medical conditions or other conditions that could affect their participation in the study such as:
* unstable angina pectoris, symptomatic congestive heart failure, myocardial infarction within 6 months of start of study drug
* serious uncontrolled cardiac arrhythmia or any other clinically significant cardiac disease
* symptomatic congestive heart failure of New York heart Association Class III or IV
* uncontrolled diabetes as defined by fasting serum glucose >1.5 x ULN
* active (acute or chronic) or uncontrolled severe infections
* liver disease such as cirrhosis, chronic active hepatitis or chronic persistent hepatitis
* A known history of HIV seropositivity
* Impairment of gastrointestinal function or gastrointestinal disease that may significantly alter the absorption of RAD001 (e.g., ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome or small bowel resection)
* Patients with an active, bleeding diathesis

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2010-02; Primary Completion 2011-06 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
To evaluate the maximum tolerated dose (MTD) and dose limiting toxicities (DLT) of RAD001 when administered in combination with chemotherapy and radiation. | 9/2011

SECONDARY OUTCOMES:
To evaluate the preliminary clinical benefit rate after administration of RAD001 in combination with chemotherapy and radiation. | 3/2012

CONTACTS AND LOCATIONS:
Overall Officials: Everett E Vokes, MD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago Medical Center, Chicago, Illinois, United States